CLINICAL TRIAL: NCT00759980
Title: Transfusing Neonates Based on Platelet Mass in the Neonatal Intensive Care Unit: A Randomized Pilot Study
Brief Title: Transfusing Neonates Based on Platelet Mass
Status: Completed | Type: Observational
Sponsor: Christiana Care Health Services (Other)
Collaborators: Alfred I. duPont Hospital for Children (Other); Thomas Jefferson University (Other); Abington Memorial Hospital (Other)
Responsible Party: Jody L. Zisk, DO, Christiana Care Health Systems
Other Study IDs: 28156
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Thrombocytopenia
Keywords: Thrombocytopenia; Platelet transfusion
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Platelet Number: Infants randomized to this group will be transfused based on a specific set of transfusion guidelines pertaining to the total number of platelets
- Platelet Mass: Infants randomized to this group will be transfused based on a specific set of transfusion guidelines pertaining to a combination of platelet number and platelet size (mass)

SUMMARY:
Thrombocytopenia (low platelet count) is common in the neonatal intensive care unit. Commonly, the decision of when to transfuse platelets is based on platelet number. Recently, Christensen et al (2006) proposed using transfusion guidelines based on platelet mass rather than platelet number. By using platelet size as a guide of when to give platelets, we may be able to decrease the amount platelet transfusions needed.

This study is investigating using platelet size rather than platelet number as a guideline for transfusing platelets in infants who are hospitalized in a NICU (neonatal intensive care unit). After obtaining parental informed consent, thrombocytopenic infants will be randomized to one of two groups. 1: Transfusion based on platelet number; 2: transfusion based on a combination of platelet number and platelet mass. In each group the decision to transfuse platelets will be made using a slightly different, yet strict set of transfusion rules.

The objective is to determine the feasibility, rate of bleeding complications and compliance of transfusing neonates based on platelet mass rather than platelet number.

The investigators hypothesize that transfusing platelets based on platelet mass will not increase bleeding complications and will reduce the number of transfusions in thrombocytopenic neonates.

ELIGIBILITY:
Inclusion Criteria:

* Thrombocytopenic infants

Exclusion Criteria:

* Major congenital anomalies

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants who are thrombocytopenic and hospitalized in the NICU
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Total number of transfusions | During NICU hospitalization

SECONDARY OUTCOMES:
Bleeding outcomes | While the infant is thrombocytopenic
Compliance with transfusion guidelines | During NICU hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Jody L Zisk, DO, Principal Investigator — Christiana Care Health Services; David A Paul, MD, Principal Investigator — Christiana Care Health Systems
Locations (4):
- United States (4):
  - Christiana Care Health System, Newark, Delaware
  - A.I. duPont Hospital for Children, Wilmington, Delaware
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania